CLINICAL TRIAL: NCT05155800
Title: A Prospective, Non-Randomized, Sequentially Enrolled, Multi-Center, Phase II Study to Evaluate the SENSE Device's Ability to Detect and Monitor Traumatic Brain Injury
Brief Title: A Study to Test the SENSE Device in Military-Age Patients With Traumatic Brain Injury
Acronym: Sense-005
Status: Completed | Type: Observational
Sponsor: Sense Diagnostics, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: Sense-005
Record Dates: First submitted 2021-11-12; First posted 2021-12-14 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (3):
- TBI patients with intracranial bleeding
  Interventions: Device: SDx3
- TBI patients without intracranial bleeding
  Interventions: Device: SDx3
- Control Subjects with normal brain health
  Interventions: Device: SDx3

INTERVENTIONS:
Device: SDx3 — The SENSE Device (SDx3) is a non-invasive device that detects differences in the absorption of transmitted RF energy across the skull and brain and is intended to be used to evaluate intracranial hemorrhage.

SUMMARY:
The study population will consist of 3 mutually-exclusive sets of patients and subjects:

* TBI patients with intracranial bleeding
* TBI patients without intracranial bleeding
* Control subjects with normal brain health.

Research subjects between the ages of 22 to 50 will be enrolled. All TBI patients must have a diagnostic head CT scan within 24 hours of the injury. TBI patients without intracranial bleeding based on the CT scan must have a Glasgow Coma Scale (GCS) score at enrollment of ≤ 14. Total maximum duration of active monitoring with the device in this study is 48 hours with a clinical follow-up at day 7 after enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet all of the following inclusion criteria will be considered candidates for study enrollment:

  * Male or female subjects age 22 to 50
  * Patients with TBI who have a diagnostic head CT scan within 24 hours of the injury.
  * For patients with TBI without intracranial hemorrhage, Glasgow Coma Scale score at enrollment of ≤ 14.
  * For patients with TBI, intended clinical monitoring in the hospital setting for at least 6 hours from study enrollment.
  * Signed written informed consent by study subject or, if subject is unable, by subject's next of kin or legal guardian.
  * Willingness and ability to comply with schedule for study procedures.
  * Control subjects with normal brain health.

Exclusion Criteria:

* All subjects meeting any of the following criteria will be excluded from this study:

  * Female patients who are pregnant or lactating.
  * Known history of seizure or clinical seizure prior to initiating SENSE monitoring.
  * Open skull fracture.
  * Metallic intracranial clip, coil, or device (such as metallic ICP monitor).
  * Presence or history of any other condition or finding that, in the investigator's opinion, makes the patient unsuitable as a candidate for the SENSE device monitoring or study participation or may confound the outcome of the study.
  * Planned placement of an intraventricular catheter after the diagnostic (pre-enrollment) CT.
  * Planned withdrawal of care within 24 hours of enrollment.
  * Planned intracranial surgery within 24 hours of enrollment.
  * Current participation in a medical or surgical interventional clinical trial.
  * Planned or current use of continuous EEG monitoring.
  * Control subjects with normal brain health will have no known history of seizure, stroke, brain tumor, TBI

Ages: 22 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of 3 mutually-exclusive sets of patients and subjects:
  * TBI patients with intracranial bleeding
  * TBI patients without intracranial bleeding
  * Control subjects with normal brain health.
  Research subjects between the ages of 22 to 50 will be enrolled. All TBI patients must have a diagnostic head CT scan within 24 hours of the injury. TBI patients without intracranial bleeding based on the CT scan must have a Glasgow Coma Scale (GCS) score at enrollment of ≤ 14.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2021-12-28 (Actual); Primary Completion 2023-10-17 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Compare ICH in TBI patients to non-ICH control subjects | up to 12 months
  1. Distinguish TBI subjects with intracranial hemorrhage from those without intracranial hemorrhage and from non-TBI controls.
Measure growth of intracranial hemorrhage | up to 12 months
  2. Detect new or enlarging intracranial hemorrhage of ≥ 6 ml among TBI subjects, as defined by CT scan.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Ratcliff, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady, Atlanta, Georgia
  - UC Health, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: Undecided
Undecided